CLINICAL TRIAL: NCT05550571
Title: Treatment of Ruptured Wide-Neck Aneurysms With Nautilus Device Assisted Occlusion
Brief Title: A Medical Device to Treat Wide-Neck Brain Aneurysms
Acronym: TORNADO-US
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EndoStream Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-329(US)
Record Dates: First submitted 2022-09-11; First posted 2022-09-22 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Ruptured Cerebral Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Patients treated with the device (Experimental)
  Interventions: Device: Nautilus Intrasaccular Bridging System

INTERVENTIONS:
Device: Nautilus Intrasaccular Bridging System — Patients will be treated with the Nautilus, then followed-up for 12 months

SUMMARY:
The study aims to evaluate the safety and probable benefit of a medical device to treat wide-neck ruptured brain aneurysms.

DETAILED DESCRIPTION:
Patients with ruptured brain aneurysms will be treated with the Nautilus, then will be followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years old
2. Subject who presents with an angiographically confirmed, wide neck intracranial saccular, acutely ruptured aneurysm. Wide neck is defined as 4-7mm.
3. Aneurysm dome ≥5 mm.
4. Subject is neurologically stable with a Hunt & Hess score of I, II, or III.
5. In the opinion of the treating physician, placement of the Nautilus is technically feasible and clinically reasonable.
6. The subject or authorized representative is able to provide informed consent and has signed the IRB-approved informed consent form.
7. Subject must be able to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule.

Exclusion Criteria:

1. Subject with any neurological deficit occurred within the last 180 days; defined as previous non-aneurysmal subarachnoid hemorrhage or any other non-aneurysmal intracranial hemorrhage, stroke, transient ischemic attacks (TIA), concussion, head trauma, cranial surgery, radiation therapy to the head.
2. Premorbid mRS score ≥3.
3. Subject has another aneurysm which, in the Investigator's opinion, will require treatment within the follow-up period (1 year).
4. Women of child-bearing potential age (18-55) who cannot provide a negative pregnancy test.
5. Subject with other serious comorbidities that carry a high risk of neurologic events such as:

   * Significant acute or chronic cardiovascular disease such as myocardial infarction within the past 180 days
   * Uncorrectable coagulation abnormality
   * Uncontrolled diabetes mellitus with target organ injury
   * Organ failure of kidney, liver, heart or lungs
   * Arteriovenous malformation or arteriovenous fistula, Moyamoya disease, or any other vasoconstriction
   * Premorbid intracranial tumor or hematoma
6. Severe or unstable conditions or diseases (e.g., non-significant neurological deficit, cancer, hematologic or coronary disease) or chronic conditions that in the opinion of the investigator may increase the risk associated with study participation for study device administration or may interfere with the interpretation of study results.
7. Extreme vessel stenosis or tortuosity or other vascular anomalies that would prevent delivery of the device to the target.
8. Comorbidities that may preclude obtaining follow-up DSA.
9. Known allergy to Nickel and/or Heparin that cannot be medically treated.
10. Subject is currently participating in another interventional clinical study.
11. Subject with a relative contraindication to angiography (i.e., allergy to contrast media, coagulopathy, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-12-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects experiencing death or stroke | 12 months
  The proportion of subjects experiencing death or stroke in treated vascular territory measured using the NIH stroke scale

SECONDARY OUTCOMES:
The proportion of subjects with complete aneurysm occlusion | 12 months
  The proportion of subjects with complete aneurysm occlusion (defined as Raymond Roy scale =1) without retreatment at 1-year follow-up imaging
device-related Serious Adverse Event | 12 months
  Proportion of subjects with a device-related Serious Adverse Event
aneurysm occlusion at the conclusion of the treatment procedure | During procedure
  Proportion of subjects with aneurysm occlusion at the conclusion of the treatment procedure (assessed via the Raymond Roy scale)
Distribution of parent vessel compromise | 12 months
  The percentage of parent vessel compromise will be evaluated by treating physician
Coil/Device entanglement | During procedure
  Proportion of events of Coil/Nautilus entanglement during implantation which precludes the coil from being removed or adjusted
Technical Success | During procedure
  Device placement success rate

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Baptist Health Ambulatory Services, Inc. d/b/a/ Baptist Health Research Institute, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - The research Foundation For The State Of New York On Behalf Of The University At Buffalo, Buffalo, New York
  - Mount Sinai, New York, New York
- UMHAT "Sv. Ivan Rilski" EAD, Sofia, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No